CLINICAL TRIAL: NCT04592822
Title: A Single Dose, Randomized, Open Label, Two-Treatment, Two-Sequence, Two-Period, Crossover Bioequivalence Study of WD-1602 Versus Pradaxa® in Healthy Subjects Under Fed Condition
Brief Title: A Single Dose Bioequivalence Study of WD-1602 Versus Pradaxa® in Healthy Subjects Under Fed Condition
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hong Kong WD Pharmaceutical Co., Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WD-1602-1001
Record Dates: First submitted 2020-10-16; First posted 2020-10-19 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Anticoagulant
MeSH Terms: interventions — Dabigatran

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment T (Experimental): 30 minutes after the start of a standard breakfast, subjects will take one straw of WD-1602 Dabigatran Etexilate Mesylate Granules (150 mg) in 100 mL water as oral administration.
  Interventions: Drug: WD-1602
- Treatment R (Active Comparator): 30 minutes after the start of a standard breakfast, subjects will receive a single Pradaxa® 150 mg capsule swallowed with 240 mL water as oral administration.
  Interventions: Drug: Pradaxa®

INTERVENTIONS:
Drug: WD-1602 — dabigatran etexilate mesylate granules for oral suspension
  Arms: Treatment T
Drug: Pradaxa® — dabigatran etexilate capsules
  Arms: Treatment R

SUMMARY:
This study will be a single-center, randomized, single-dose, open-label, two-treatment, two-period, two-sequence crossover bioequivalence study to compare the rate and extent of absorption of WD-1602 granule formulation (WD Pharma) to the reference drug Pradaxa® capsule (BI, Germany) under fed conditions in healthy subjects.

DETAILED DESCRIPTION:
The study will comprise of a medical Screening visit, two 2-night (3-day) Treatment Periods, 2 outpatient visits, and a Follow-up visit. Each Treatment visit will be separated by a washout of up to 7 days. The Follow-up visit will occur approximately 7 days (±1) following the last study drug administration. The duration of subject participation, including screening, will be approximately 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria: based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead; electrocardiogram (ECG), clinical laboratory tests.
2. Ages of 18 and 55 years, inclusive, who have a minimum body weight of 50.0 kg (110.0 lbs.) and ≤ 100 kg (220 lbs.).
3. Body Mass Index (BMI) between 18.0 and 29.0 kg/m2, inclusive.
4. Negative urine pregnancy test in women of childbearing potential who are not actively breastfeeding, do not plan to become pregnant during the study, and agree to use an approved method of birth control (abstinence from heterosexual activity that could result in conception, hormonal contraceptives, condom with spermicide, diaphragm or cervical cap with spermicide, or intrauterine device) for the duration of study participation; or women of nonchildbearing potential who are > 1 year postmenopausal with follicle-stimulating hormone in the postmenopausal range.
5. Willingness of male subjects to use barrier contraception (condom with spermicide) and refrain from donating sperm, for the duration of study participation.
6. Normal coagulation function (prothrombin time [PT] and partial thromboplastin time [PTT] < 1.2 x upper limit of normal of normal [ULN] laboratory reference range).
7. Normal hepatic function (alanine aminotransferase [ALT] < 1.2 × ULN; total bilirubin level < 2 × ULN).
8. Normal renal function (estimated glomerular filtration rate > 60 mL/min/1.73 m2).
9. Ability to understand informed consent, which must be signed before any study-related procedures are performed in accordance with Good Clinical Practice (GCP) and the local legislation.

Exclusion Criteria:

1. Clinically significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders.
2. Clinically significant surgery of gastrointestinal tract or evidence of significant gastrointestinal motility problems that could affect absorption of the drug.
3. Diseases of the central nervous system (included but not limited to any kind of seizures; stroke or psychiatric disorders).
4. Any history or evidence of blood dyscrasia, hemorrhagic diathesis, severe thrombocytopenia, cerebrovascular hemorrhage, bleeding tendencies associated with active ulceration or overt bleeding of gastrointestinal, respiratory or genitourinary tract or any disease or condition with hemorrhagic tendencies.
5. History of significant orthostatic hypotension, fainting spells or blackouts.
6. Chronic or relevant acute infections.
7. History of allergy/hypersensitivity (including drug allergy in particular to study drug or its excipients) which is deemed relevant to the trial as judged by the Principal Investigator (i.e., an Ontario-licensed physician) or Sub-Investigator (Ontario-licensed physician and/or Nurse Practitioner)..
8. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial.
9. Alcohol abuse (more than 20 g/day).
10. Drug abuse.
11. Blood donation (more than 100 mL within four weeks prior to administration or during the trial);
12. Participation in another trial with an investigational drug within four weeks prior to administration or during the trial.
13. Any laboratory value outside the reference range that is of clinical significance or positive drug or virus screening.
14. Planned surgeries within four weeks following the end-of study examination; and
15. Recent or contemplated diagnostic or therapeutic procedures with potential for uncontrollable bleeding within days before or after end-of study examination.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-06 (Estimated); Primary Completion 2021-06-06 (Estimated); Study Completion 2021-12-06 (Estimated)

PRIMARY OUTCOMES:
AUC0-t | pre-dose (baseline) and day 1, day 2, day 3 post-dose at designed time intervals.
  area under the plasma concentration-time curve from time 0 to time t
AUC0-inf | pre-dose (baseline) and day 1, day 2, day 3 post-dose at designed time intervals.
  area under the concentration-time curve from time 0 to time infinity
Cmax | pre-dose (baseline) and day 1, day 2, day 3 post-dose at designed time intervals.
  the maximum concentration